CLINICAL TRIAL: NCT00506948
Title: Thymoglobulin, Sirolimus and Mycophenolate Mofetil for Prevention of Acute GVHD Following Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Thymoglobulin, Sirolimus and Mycophenolate Mofetil for Prevention of Acute Graft-Versus-Host Disease (GVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to high incidence of veno-oclusive disease of the liver.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0435
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2014-02-20 (Estimated); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Hematological Malignancies; Myelodysplastic Syndrome; Leukemia; Lymphoma
Keywords: Hematological Malignancies; Myelodysplastic Syndrome; Graft Versus Host Disease; GVHD; Allogeneic Hematopoietic Stem Cell Transplantation; AHSCT; Leukemia; Lymphoma; T-Cells; Thymoglobulin; ATG; rATG; Rabbit Antithymocyte Globulin; Rapamune; Sirolimus; Mycophenolate Mofetil; Cellcept; MMF
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia; Lymphoma; Graft vs Host Disease | interventions — Mycophenolic Acid; thymoglobulin; Antilymphocyte Serum; Sirolimus; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thymoglobulin + Sirolimus + MMF (Experimental): Thymoglobulin 1.5 mg/kg intravenous (IV) days -4, -3, -2, -1 before Stem Cell Transplant (Day 0); Sirolimus 6 mg IV on day -2 followed by 2 mg daily to maintain therapeutic levels and Mycophenolate Mofetil (MMF) 15 mg/kg IV or orally every 12 hours starting on day 0 until day+27.
  Interventions: Drug: Mycophenolate Mofetil (MMF); Drug: Thymoglobulin; Drug: Sirolimus; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Mycophenolate Mofetil (MMF) — 15 mg/kg by vein or by mouth every 12 hours.
  Other Names: CellCept; MMF
Drug: Thymoglobulin — 1.5 mg/kg by vein daily for 4 days
  Other Names: Antithymocyte Globulin; rATG; ATG
Drug: Sirolimus — 6 mg daily by mouth for 1 day, followed by 2 mg daily for 1 day.
  Other Names: Rapamune
Procedure: Stem Cell Transplant — Stem cell infusion on Day 0.
  Other Names: hematopoietic stem cell transplantation; HSCT; transplantation

SUMMARY:
The goal of this clinical research study is to learn if the combination of rabbit anti-thymocyte globulin (Thymoglobulin®), sirolimus (Rapamune®), and mycophenolate mofetil (Cellcept®) can help to prevent graft versus host disease (GVHD). The safety of this drug combination will also be studied.

Primary Objective: To determine efficacy and toxicity of a regimen of thymoglobulin, sirolimus and mycophenolate mofetil for prevention of acute GVHD after allogeneic stem cell transplantation from human leukocyte antigen (HLA) identical related or unrelated donors.

Secondary Objective: To assess engraftment, chronic GVHD, relapse and survival.

DETAILED DESCRIPTION:
Rabbit anti-thymocyte globulin (rATG), sirolimus, and mycophenolate mofetil (MMF) are all designed to prevent GVHD.

If you are found to be eligible to take part in this study, you will receive rATG through a needle in your vein over 3-4 hours on each of the 4 days before the stem cell transplant.

Beginning 2 days before the transplant, you will take sirolimus by mouth once per day. You will continue to receive sirolimus until 90 days after the transplant. Beginning on Day 60, you will start taking increasingly lower doses of the study drug. This is done so you can taper down slowly, and be off of the drug on Day 90.

Beginning on the day of the transplant, you will take MMF by mouth 2 times a day. You will continue to take MMF until 27 days after the transplant.

Every week (for the first 90-100 days after the transplant) you will have study visits. At this visit, you will have a physical exam. Blood (about 1-2 tablespoons) will be drawn for routine tests.

You will remain on study for up to 90 days after transplantation. You will be taken off study if intolerable side effects occur.

Starting on Day 90 after the transplant, you will continue to follow up with your transplant doctor at least every 3 months through 1 year after the transplant. During these visits you will have physical exams. Blood (about 1-2 tablespoons) will be drawn for routine tests. Your doctor may request additional testing.

This is an investigational study. RATG, sirolimus, and MMF are all FDA approved for their use in the transplantation of solid organs (like kidney and liver). All 3 drugs are commercially available. This particular combination and dose schedule is considered investigational. Up to 30 patients will take part in this study. All will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high risk hematological malignancies, including those with induction failure and after treated or untreated relapse. High risk hematological malignancies include: Acute myelogenous or lymphocytic leukemia with induction failure of after relapse, myelodysplastic syndrome of intermediate and high risk according to Greenberg criteria, chronic myelogenous leukemia in accelerated phase or blast crisis, non-Hodgkin's and Hodgkin's lymphoma with induction failure or relapse after chemotherapy and refractory or relapsed chronic lymphocytic leukemia.
2. HLA-identical sibling or matched unrelated donor transplants not eligible for protocols of higher priority.
3. Age 18-75 years.
4. Bilirubin </=1.5 mg/dl, serum glutamic-pyruvic transaminase (SGPT) </= 200 IU/ml.
5. Creatinine </=1.6 mg/dl.

Exclusion Criteria:

1. Regimens including rituximab or alemtuzumab in the preparative regimen.
2. Patients can not have received prior treatment with gemtuzumab.
3. Planned conditioning chemotherapy for transplant can not include gemtuzumab.
4. Planned conditioning chemotherapy for transplant can not include the busulfan and cyclophosphamide regimen.
5. HIV seropositivity
6. Uncontrolled infection, not responding to adequate antimicrobial therapy after 7 days of treatment. The protocol PI is the final arbiter of eligibility.
7. Pregnancy
8. Inability to sign consent.
9. Patients who are past recipients of allogeneic or autologous stem cell transplants from any source.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 08, 2006 to October 27, 2009. All recruitment done in a medical clinic setting.
Pre-assignment Details: Of the 13 participants enrolled, three participants were ineligible and excluded from the study before treatment.
Period: Overall Study
Arm/Group | Thymoglobulin + Sirolimus + MMF
Started | 10
Completed | 0
Not Completed | 10
Not completed — Death | 4
Not completed — Adverse Event | 5
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thymoglobulin + Sirolimus + MMF
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Failure Rate
Description: Efficacy failure defined as a participants who had either grade 3-4 acute graft-versus-host disease (aGVHD) or treatment related mortality (TRM) within 100 days post transplant. Failure Rate calculated as (# of failures) / (# participants evaluated). Physical exam and bloodwork every week (for the first 90-100 days after the transplant).
Time Frame: Baseline to 100 days post transplant
Reporting Status: Not Posted

2. Primary Outcome: Number of Participants With Acute Graft-versus-host Disease (aGVHD)
Description: Participants who had acute graft-versus-host disease (aGVHD) within 100 days post transplant. Physical exam and bloodwork every week (for the first 90-100 days after the transplant).
Time Frame: Baseline to 100 days post transplant
Measure: Number; unit: participants
Arm/Group | Thymoglobulin + Sirolimus + MMF
Number analyzed (Participants) | 10
participants | 6

ADVERSE EVENTS:
Time Frame: Adverse event reporting from active treatment completed on day 90 (last day of sirolimus) through post-study surveillance to Day +100. Adverse events were collected for a total study period of 2 years and 11 months.
Arm/Group | Thymoglobulin + Sirolimus + MMF
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin + Sirolimus + MMF (N=10)
Death (General disorders) | 4 — Two deaths related to cases of veno-occlusive disease of the liver.
Veno-occlusive disease of the liver (Renal and urinary disorders) | 4 — Two of the four cases were fatal.
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Thymoglobulin + Sirolimus + MMF (N=10)
Nausea (Gastrointestinal disorders) | 2 — Grade 2
Hemorrhagic Cystitis (Renal and urinary disorders) | 1
Veno-occlusive disease of the liver (Moderate) (Renal and urinary disorders) | 2
Skin GVHD (Skin and subcutaneous tissue disorders) | 2
Gastrointestinal GVHD (Gastrointestinal disorders) | 2
Acute GVHD (General disorders) | 2 — Liver, skin (rash), mucosa, and gastrointestinal tract.

LIMITATIONS AND CAVEATS:
A decision to terminate this trial was made due to the high incidence of veno-occlusive disease of the liver in participants receiving this graft-versus-host disease (GVHD) prophylaxis regimen.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No